CLINICAL TRIAL: NCT01229410
Title: Pharmacokinetics of the Brimonidine Tartrate Posterior Segment Delivery System in Patients Undergoing Pars Plana Vitrectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 190342-036
Record Dates: First submitted 2010-10-20; First posted 2010-10-27 (Estimated); Results first posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-07

CONDITIONS: Vitrectomy
MeSH Terms: interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 400 µg Brimonidine Tartrate Implant (Experimental): 400 µg brimonidine tartrate implant in the study eye on Day 1 (2, 4 or 8 weeks prior to undergoing a pars plana vitrectomy).
  Interventions: Drug: 400 µg Brimonidine Tartrate Implant
- 200 µg Brimonidine Tartrate Implant (Experimental): 200 µg brimonidine tartrate implant in the study eye on Day 1 (2, 4 or 8 weeks prior to undergoing a pars plana vitrectomy).
  Interventions: Drug: 200 µg Brimonidine Tartrate Implant

INTERVENTIONS:
Drug: 400 µg Brimonidine Tartrate Implant — 400 µg brimonidine tartrate implant in the study eye on Day 1 (2, 4 or 8 weeks prior to undergoing a pars plana vitrectomy).
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 400 µg Brimonidine Tartrate Implant
Drug: 200 µg Brimonidine Tartrate Implant — 200 µg brimonidine tartrate implant in the study eye on Day 1 (2, 4 or 8 weeks prior to undergoing a pars plana vitrectomy).
  Other Names: Brimonidine Tartrate PS DDS®
  Arms: 200 µg Brimonidine Tartrate Implant

SUMMARY:
This study will evaluate the pharmacokinetics of brimonidine following a single intravitreal administration of the 200 ug or 400 ug Brimonidine Tartrate Posterior Segment Drug Delivery System in patients 2, 4 or 8 weeks prior to undergoing a pars plana vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Plan on having a pars plana vitrectomy for repair of a posterior segment condition (eg, epiretinal membrane, macular hole, vitreomacular traction)
* Visual acuity in the non-study eye better than 20/200

Exclusion Criteria:

* History of pars plana vitrectomy or retinal detachment surgery in the study eye
* Surgery or laser treatment in the study eye within 3 months
* Use of brimonidine, apraclonidine or other topical alpha-2-agonist in either eye within 2 weeks
* Intraocular infection or inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Salt Lake City, Utah, United States
- Prague, Czechia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were enrolled in groups by planned time of pars plana vitrectomy (Week 2, 4, or 8 post-implant). Patients who had the implant removed during the vitrectomy did not complete the 6 month follow-up per protocol.
Period: Overall Study
Arm/Group | 400 µg Brimonidine Tartrate Implant | 200 µg Brimonidine Tartrate Implant
Started | 12 | 12
Completed | 7 | 9
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 400 µg Brimonidine Tartrate Implant | 200 µg Brimonidine Tartrate Implant | Total
Number analyzed (Participants) | 12 | 12 | 24
Age Continuous [Mean (Full Range); unit: Years] | 69.7 (2.87) [64 to 75] | 66.5 (9.67) [53 to 78] | 68.1 [53 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Highest Vitreous Humor Level of Brimonidine in the Study Eye
Description: The highest level of brimonidine measured in the vitreous humor of the study eye in any patient is reported for each treatment arm. The vitreous humor is the clear gel that fills the space between the lens and the retina of the eye.
Time Frame: 60 Days
Population: Per Protocol: all subjects with pharmacokinetic data available
Measure: Number; unit: Nanogram/milliliter (ng/mL)
Arm/Group | 400 µg Brimonidine Tartrate Implant | 200 µg Brimonidine Tartrate Implant
Number analyzed (Participants) | 11 | 12
Nanogram/milliliter (ng/mL) | 137.0 | 34.9

2. Secondary Outcome: Highest Aqueous Humor Level of Brimonidine in the Study Eye
Description: The highest level of brimonidine measured in the aqueous humor of the study eye in any patient is reported for each treatment arm. The aqueous humor is the clear fluid in the chamber of the eye between the cornea and the lens.
Time Frame: 60 Days
Population: Per Protocol: all subjects with pharmacokinetic data available
Measure: Number; unit: Nanogram/milliliter (ng/mL)
Arm/Group | 400 µg Brimonidine Tartrate Implant | 200 µg Brimonidine Tartrate Implant
Number analyzed (Participants) | 12 | 10
Nanogram/milliliter (ng/mL) | 17.5 | 12.5

3. Secondary Outcome: Percentage of Patient Samples With Plasma Levels of Brimonidine Below the Limit of Quantitation (BLQ)
Description: Percentage of patient samples with plasma levels of brimonidine reported as BLQ (i.e., too low to be determined using standard methods). Plasma is the fluid portion of the blood.
Time Frame: 60 Days
Population: Per Protocol: all subjects with qualified pharmacokinetic samples
Measure: Number; unit: Percentage of Patient Samples
Units Other Than Participants: Patient Samples
Arm/Group | 400 µg Brimonidine Tartrate Implant | 200 µg Brimonidine Tartrate Implant
Number analyzed (Participants) | 11 | 11
Number analyzed (Patient Samples) | 60 | 62
Percentage of Patient Samples | 53.3 | 72.6

ADVERSE EVENTS:
Description: For Ocular AEs, only those occurring in the study eye are reported in the "Other Adverse Events" section. For SAEs, all ocular events are reported, regardless of the eye.
Arm/Group | 400 µg Brimonidine Tartrate Implant | 200 µg Brimonidine Tartrate Implant
Serious Adverse Events (participants affected / at risk) | 1/12 | 2/12
Other Adverse Events (participants affected / at risk) | 11/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 400 µg Brimonidine Tartrate Implant (N=12) | 200 µg Brimonidine Tartrate Implant (N=12)
Choroidal Detachment (Eye disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Vitreous Haemorrhage (Eye disorders) | 0 | 1
Retinal Detachment (Eye disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 400 µg Brimonidine Tartrate Implant (N=12) | 200 µg Brimonidine Tartrate Implant (N=12)
Conjunctival Haemorrhage (Eye disorders) | 7 | 6
Conjunctival Hyperaemia (Eye disorders) | 5 | 7
Conjunctival Oedema (Eye disorders) | 2 | 2
Hypertension (Vascular disorders) | 2 | 0
Intraocular Pressure Increased (Investigations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 1 | 1
Cataract (Eye disorders) | 1 | 1
Eye Pain (Eye disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Cataract Nuclear (Eye disorders) | 1 | 0
Choroidal Detachment (Eye disorders) | 1 | 0
Hypotony of Eye (Eye disorders) | 1 | 0
Phlebitis Superficial (Vascular disorders) | 1 | 0
Vitreous Haemorrhage (Eye disorders) | 0 | 2
Retinal Detachment (Eye disorders) | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Device Dislocation (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Visual Acuity Reduced (Eye disorders) | 0 | 1
Chorioretinal Disorder (Eye disorders) | 0 | 1
Eyelid Oedema (Eye disorders) | 0 | 1
Intraocular Pressure Decreased (Investigations) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Retinal Tear (Eye disorders) | 0 | 1
Retinopathy Proliferative (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.